CLINICAL TRIAL: NCT00427375
Title: Phase III Randomized Trial of Local Excision Versus Total Mesorectal Excision in Downstaged T2T3 Low Rectal Cancer After Radiochemotherapy
Brief Title: Local Excision in Downstaged Rectal Cancer
Acronym: GRECCAR 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Sanofi (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2006/03; 2005-025
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Rectal Neoplasms
Keywords: Rectal cancer surgery; Neoadjuvant radiochemotherapy; Randomized clinical trial; Multicenter study
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): New surgical option in good responders after neoadjuvant treatment for low rectal cancer
  Interventions: Procedure: local rectal excision
- 2 (Active Comparator): Standard surgery
  Interventions: Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: local rectal excision — New surgical option in good responders after neoadjuvant treatment for low rectal cancer
  Arms: 1
Procedure: total mesorectal excision — standard surgery
  Arms: 2

SUMMARY:
Patients with T2T3 low rectal cancer (size =< 4 cm) received neoadjuvant treatment (50Gy in 5 weeks with concomitant chemotherapy. Good responders (residual tumour =< 2 cm) are randomised in local vs rectal excision, 6-8 weeks after treatment. The composite end point evaluates the rate of patients with death, recurrence, major morbidity or severe after effects at two years.

DETAILED DESCRIPTION:
Rectal excision is the standard surgical treatment of rectal cancer. The risk of mortality and major short and long term morbidity induced by rectal excision justifies new treatments. Local excision is a conservative alternative approach associated with low mortality and morbidity. The purpose of this prospective randomised multicenter study is to compare local vs rectal excision in good responders after radiochemotherapy for low rectal cancer.

Patients with T2T3 low rectal cancer, less than 8 cm from the anal verge, size =< 4 cm, received neoadjuvant treatment, included radiotherapy between 45-55Gy in 5 weeks with concomitant chemotherapy consist of at least, one fluoropyrimidine.

Good clinical responders (residual tumour =< 2 cm) are randomised in local vs rectal excision, 6-8 weeks after treatment. In case of not confirmed pathological response following local excision, complementary rectal excision is required.

Bad responders (residual tumour > 2cm) are treated by primary rectal excision. Follow-up includes digital rectal examination, CT-scan and endorectal ultrasound (if local excision) every 4 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* T2T3 low adenocarcinoma of the rectum
* Tumour size =< 4cm
* Less than 8 cm from the anal verge
* No metastatic disease
* Patient is at least 18 years of age
* ECOG performance status score =< 2
* Patient and doctor have signed informed consent
* inclusion criteria : Residual clinical tumour size =< 2cm after radiochemotherapy

Exclusion Criteria:

* T1, T4 tumour or anal sphincter invasion
* Metastatic disease (M1)
* Contra indication for radiotherapy and/or fluoropyrimidine use in chemotherapy
* History of cancer
* Symptomatic cardiac or coronary insufficiency
* Severe renal insufficiency
* Peripheral neuropathy
* Patient included in a trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-03-05 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients presenting at least 1 component of the composite outcome (4 components: death, recurrence, major morbidity and severe after effects) at 2 years after | 24 months

SECONDARY OUTCOMES:
Compare the incidence at 2 years of each component separately: death, recurrence, major morbidity and severe after effect | 24 months
5-year survival. | 5 years
Quality of life (QLQ C30 - CR38) | at 0, 4, 8 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric RULLIER, Pr., Principal Investigator — University Hospital, Bordeaux
Locations (40):
- France (40):
  - Centre Radiothérapie Oncologie Moyenne Garonne - 13 Quai du Docteur Calabet, Agen
  - Polyclinique Sainte marguerite, Auxerre
  - Service de Chirurgie Viscérale, Digestive et Cancérologique - CHRU J.Minoz - Boulevard Fleming, Besançon
  - Service de Radiothérapie - Clinique Tivoli - 220 rue Mandron, Bordeaux
  - Service de chirurgie digestive - hôpital Saint André - 1 rue Jean Burguet, Bordeaux
  - Service de Chirurgie Oncologique - Institut Bergonié - 229, cours de l'Argonne, Bordeaux
  - Service de Chirurgie Digestive - Hôpital ambroise Paré - 9 avenue Charles de Gaulle, Boulogne-Billancourt
  - Service de Chirurgie Générale et Digestive - Hôtel Dieu - CHU Clermont-Ferrand - Boulevard Léon Malfreyt, Clermont-Ferrand
  - Département de Radiothérapie - Centre Jean Perrin - 58 rue Montalembert, Clermont-Ferrand
  - Service de Chirurgie Générale et Digestive - Hôpital Beaujon - 100 boulevard du Général Leclerc, Clichy
  - Centre d'Oncologie et Radiothérapie - rue du Dr Schweitzer, La Rochelle
  - Service de Chirurgie Digestive - Hôpital A. Michallon - CHU de Grenoble - Boulevard de la Chantourne, La Tronche
  - Département de Chirurgie Oncologique - Centre Oscar Lambret - 3 rue Combemale, Lille
  - Service de Chirurgie Générale - Hôpitaux Civils de Lyon, Lyon
  - Département de Chirurgie Oncologique - Centre Léon Bérard - 28 rue Laennec, Lyon
  - Institut Paoli Calmette, Marseille
  - Service de Chirurgie Digestive et viscérale - CHU Timone - 264 rue Saint Pierre, Marseille
  - Département de Chirurgie Oncologique - CRLC Val d'Aurelle, Montpellier
  - CHU Nantes, Nantes
  - Service d'Oncologie-Radiothérapie - Centre antoine Lacassagne - 33 avenue de Valombrose, Nice
  - Service de Chirurgie Générale - Hôpital Archet II, Nice
  - CHU Nîmes, Nîmes
  - Département Médico-Chirurgical de Pathologie Digestive - Hôpital Lariboisière - 2 rue Ambroise Paré, Paris
  - Service de Cancérologie - Radiothérapie - Hôpital Saint-Louis - 1 avenue Claude Vellefeaux, Paris
  - Service de Chirurgie Digestive - Hôpital des Diaconnesses - la Croix Saint-Simon - 125 rue d'Avron, Paris
  - Service de Chirurgie Générale et Digestive - Hôpital Saint-Antoine - 184 rue du Faubourg Saint-Antoine, Paris
  - Service d'Oncologie - Radiothérapie - Hôpital Tenon - 4 rue de la Chine, Paris
  - Service de Radiothérapie - Oncologie - Centre Hospitalier Lyon Sud - Hôpitaux Civils de Lyon - 165 chemin du Grand Revoyet, Pierre-Bénite
  - Service de Chirurgie Viscérale - CHU pontchaillou - 2 rue Henri Le Guilloux, Rennes
  - Département des Radiations - Centre Eugène Marquis - rue de la Bataille Flandres-Dunkerque, Rennes
  - Service de Chirurgie Digestive - CHU Charles Nicolle - 1 rue Germont, Rouen
  - Service de Radiothérapie-Oncologie - centre Henri Becquerel - rue d'Amiens, Rouen
  - Service de Chirurgie Oncologique - Centre René Gauducheau - Boulevard Jacques Monod, Saint-Herblain
  - Service de Chirurgie Viscérale - Clinique Charcot - 51-52 rue Commandant Charcot, Sainte-Foy-lès-Lyon
  - Département de Radiothérapie - Centre Paul Strauss - 3 rue de la Porte de l'Hôpital, Strasbourg
  - Service de Chirurgie Digestive - Hôpital Hautepierre, Strasbourg
  - Département d'Oncologie Médicale - Institut Claudius Régaud - 20-24 rue du Pont Saint Pierre, Toulouse
  - Service de Chirurgie Digestive - Hôpital Purpan - Place du Docteur Baylac, Toulouse
  - Département de Chirurgie Oncologique - Centre Alexis Vautrin - Avenue de Bourgogne, Vandœuvre-lès-Nancy
  - Service de Chirurgie Digestive et Générale - CHU Brabois - avenue de Bourgogne, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teste B, Rouanet P, Tuech JJ, Valverde A, Lelong B, Rivoire M, Faucheron JL, Jafari M, Portier G, Meunier B, Sielezneff I, Prudhomme M, Marchal F, Dubois A, Capdepont M, Denost Q, Rullier E. Early and late morbidity of local excision after chemoradiotherapy for rectal cancer. BJS Open. 2021 May 7;5(3):zrab043. doi: 10.1093/bjsopen/zrab043. PMID 34097005
- [Derived] Rullier E, Vendrely V, Asselineau J, Rouanet P, Tuech JJ, Valverde A, de Chaisemartin C, Rivoire M, Trilling B, Jafari M, Portier G, Meunier B, Sieleznieff I, Bertrand M, Marchal F, Dubois A, Pocard M, Rullier A, Smith D, Frulio N, Frison E, Denost Q. Organ preservation with chemoradiotherapy plus local excision for rectal cancer: 5-year results of the GRECCAR 2 randomised trial. Lancet Gastroenterol Hepatol. 2020 May;5(5):465-474. doi: 10.1016/S2468-1253(19)30410-8. Epub 2020 Feb 7. PMID 32043980
- [Derived] Rullier E, Rouanet P, Tuech JJ, Valverde A, Lelong B, Rivoire M, Faucheron JL, Jafari M, Portier G, Meunier B, Sileznieff I, Prudhomme M, Marchal F, Pocard M, Pezet D, Rullier A, Vendrely V, Denost Q, Asselineau J, Doussau A. Organ preservation for rectal cancer (GRECCAR 2): a prospective, randomised, open-label, multicentre, phase 3 trial. Lancet. 2017 Jul 29;390(10093):469-479. doi: 10.1016/S0140-6736(17)31056-5. Epub 2017 Jun 7. PMID 28601342